CLINICAL TRIAL: NCT04991519
Title: Understanding the Brain Basis of Language and Cognitive Functions Through the Study of Individuals With Brain Injury and Healthy Controls
Brief Title: Brain-based Understanding of Individual Language Differences After Stroke
Acronym: BUILD
Status: Active, not recruiting | Type: Observational
Sponsor: Georgetown University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Drexel University (Other); MedStar National Rehabilitation Network (Other)
Responsible Party: Sponsor
Other Study IDs: BUILD; R01DC014960 (NIH)
Record Dates: First submitted 2021-07-01; First posted 2021-08-05 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-04

CONDITIONS: Aphasia; Stroke; Alexia
Keywords: aphasia; stroke; brain injury; speech; language; reading; alexia; apraxia
MeSH Terms: conditions — Aphasia; Stroke; Dyslexia; Brain Injuries; Speech; Language; Apraxias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke Survivors: Participants have had a left-hemisphere stroke with or without aphasia, or a stroke elsewhere in the brain causing aphasia. They are given a series of standardized and in-house tests of language and cognition to provide a detailed profile of strengths and weaknesses, plus an MRI.
- Controls: Participants are matched to aphasia cohort in age, educational background, race, and gender but have no history of brain injury. They are also given a series of standardized and in-house tests of language and cognition to provide a detailed profile of strengths and weaknesses, plus an MRI.

SUMMARY:
Strokes often cause a loss of communication ability, referred to as aphasia, as well as cognitive difficulties. Each stroke survivor has a unique pattern of strengths and weaknesses in communication and cognition, and a unique course of recovery. The BUILD study aims to understand the brain basis of these individual differences in stroke outcome. Participants with stroke as well as controls matched in age, educational background, race, and sex are examined using a combination of standardized and in-house tests of language and cognition to provide a detailed profile of strengths and weaknesses. Each participant will have between three and six sessions, including an MRI to measure details of the structure, function, and connections in the brain. The data are analyzed to test how patterns in the stroke lesion explain the patterns of communication and cognitive difficulties, and how patterns in the uninjured parts of the brain explain resilience and recovery from the stroke. Ultimately, we hope that BUILD will guide us toward new targets for brain stimulation treatments or other biologically based treatments that improve language and cognitive abilities after stroke.

ELIGIBILITY:
Inclusion Criteria:

Stroke Survivors:

* Age >=18
* Stroke in left hemisphere of brain with or without aphasia, or stroke elsewhere causing aphasia
* Learned English at 8 years or younger

Controls:

* Age >=18
* No history of brain injury resulting from stroke, trauma, infection (i.e. encephalitis), or tumor
* Learned English at 8 years or younger

Exclusion Criteria:

* History of other brain conditions that could impact interpretation of results (such as multiple sclerosis, premorbid dementia)
* Severe psychiatric condition that would interfere with participation in the study
* History of a learning disability that could impact interpretation of results

Additional Exclusion Criteria for MRIs:

* Pacemaker or magnetic metal in the body that is not MRI compatible
* Pregnancy
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are survivors of left hemisphere stroke with or without aphasia, or people with aphasia due to strokes in other parts of the brain. We recruit participants primarily from the Washington, DC region, but some participants may travel from farther away to participate in the study. We aim for our participants to be fully representative of the diversity of individuals with stroke in the general population. Control participants are matched to stroke survivors on age, gender, race, educational background, and stroke risk factors.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
MP-RAGE (Magnetization Prepared Rapid Acquisition Gradient Echo) | Collected within 1 month of behavioral testing
  Part of MRI sequence that measures deep grey matter structure.
DTI (Diffusion Tensor Imaging) | Collected within 1 month of behavioral testing
  Part of MRI sequence that measures the rate of water diffusion between cells to understand and create a map of internal structures.
Behavioral testing | Collected within 1 month of MRI
  Battery of standard clinical and in-house behavioral tests to measure speech, language, and cognition. Final score is derived from principle components analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Turkeltaub, MD,PhD, Principal Investigator — Georgetown University; MedStar National Rehabilitation Hospital
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

DOCUMENTS (1):
  • Study Protocol (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT04991519/Prot_000.pdf